CLINICAL TRIAL: NCT03486678
Title: A Single-arm, Open-label and Exploratory Clinical Study of PD-1 Monoclonal Antibody SHR-1210 in Combination With GEMOX (Gemcitabine Combined Oxaliplatin) in Patients With Advanced Biliary Tract Cancer
Brief Title: SHR-1210 in Combination With GEMOX in Patients With Advanced BTC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR1210-GEMOX-BTC-IIT03
Record Dates: First submitted 2018-02-01; First posted 2018-04-03 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Biliary Tract Cancer; Cholangiocarcinoma
Keywords: BTC; PD-1 antibody
MeSH Terms: conditions — Biliary Tract Neoplasms; Cholangiocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR1210+GEMOX (Experimental): This is a single arm trial. Participants will receive SHR1210 + GEMOX treatment.
  Interventions: Drug: SHR-1210+GEMOX

INTERVENTIONS:
Drug: SHR-1210+GEMOX — 28 days as a treatment cycle, SHR-1210 3mg/kg and Gemcitabine 800 mg/m2 will be administered IV Q2W (D1 and D15 of a treatment cycle),and Oxaliplatin 85mg/m2 will be administered IV Q2W (D2 and D16 of a treatment cycle). PD-1 antibody combined chemotherapy used up to 6 cycles.SHR-1210 3mg/kg IV Q2W will be administered beyond chemotherapy until the disease progression or untolerable toxicity.

SUMMARY:
This is a single-arm, open-label and exploratory clinical study of PD-1 monoclonal antibody SHR-1210 combined with GEMOX regimen (gemcitabine combined oxaliplatin) in the treatment of advanced biliary malignancies.

In oder to observe and evaluate the efficacy and safety of PD-1 antibody SHR-1210 combined with GEMOX in the treatment of patients with advanced biliary malignant tumor (BTC),subjects with pathological confirmed biliary cancer, including intrahepatic bile duct carcinoma, extrahepatic bile duct carcinoma, and gallbladder carcinoma will be enrolled.

28 days as a treatment cycle, SHR-1210 3mg/kg and Gemcitabine 800 mg/m2 will be administered IV Q2W (D1 and D15 of a treatment cycle),and Oxaliplatin 85mg/m2 will be administered IV Q2W (D2 and D16 of a treatment cycle). PD-1 antibody combined chemotherapy will be used up to 6 cycles.SHR-1210 3mg/kg IV Q2W will be administered beyond 6 cycles chemotherapy until disease progression or un-tolerable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Pathology confirmed biliary malignancy, including intrahepatic bile duct carcinoma, extrahepatic bile duct carcinoma, and gallbladder carcinoma.
* Age:18-75 years, male or female.
* The estimated survival period is more than 3 months.
* ECOG 0-1.
* There is at least one measurable lesion, according to the RECIST 1.1 standard.
* Patients has not been treated by oxaliplatin, gemcitabine and pd-1 / pd-l1 antibody.
* Patients who have been treated tegafur or capecitabine as adjuvant chemotherapy or first-line treatment may be selected.

Exclusion Criteria:

* There were concurrent malignant tumors, except for the cured skin basal cell carcinoma and cervical carcinoma in situ.
* Other drug clinical trials have been taken in four weeks.
* Patients with a history of central nervous system metastasis or central nervous system metastasis are known before the screening.
* Patients with a history of unstable angina.
* The urine routine indicated that the urine protein was greater than ++ and confirmed the 24-hour urine protein quantification >1.0 g.
* Have used immune-targeted therapy drugs.
* The patient had received a liver transplant.
* Having a history of chronic autoimmune diseases such as systemic lupus erythematosus.
* Having a history of immunodeficiency, or other acquired, congenital immunodeficiency diseases, or a history of organ transplantation;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2018-02-10 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
6-month Progression Free Survival (PFS) rate | from the first drug administration up to 6 months
  the rate of 6-month progression free survival
Incidence of Treatment-Emergent Adverse Events | from the first drug administration to within 90 days for the last SHR-1210 dose
  Incidence of Treatment-Emergent Adverse Events, especially immune related adverse events

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | from the first drug administration up to two years
  the best Objective Response Rate
Duration of response (DOR) | from the first drug administration up to two years
  Duration of response
Disease Control Rate (DCR) | from the first drug administration up to two years
  the Rate of Disease Control
12-month Overall survival (OS) rate | from the first drug administration up to approximately 12 months
  Overall Survival rate at 12 months
OS | from the first drug administration up to 2 years
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Yongqian Shu, PhD, Principal Investigator — JANGSU PROVINCE HOSPITAL
Locations (1):
- Jiangsu Province Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu QP, Tang J, Chen YZ, Guo F, Ma L, Pan LL, Tian YT, Wu XF, Zhang YD, Chen XF. Immuno-genomic-radiomics to predict response of biliary tract cancer to camrelizumab plus GEMOX in a single-arm phase II trial. JHEP Rep. 2023 Apr 22;5(7):100763. doi: 10.1016/j.jhepr.2023.100763. eCollection 2023 Jul. PMID 37333974
- [Derived] Chen X, Wang D, Liu J, Qiu J, Zhou J, Ying J, Shi Y, Wang Z, Lou H, Cui J, Zhang J, Liu Y, Zhao F, Pan L, Zhao J, Zhu D, Chen S, Li X, Li X, Zhu L, Shao Y, Shu Y. Genomic alterations in biliary tract cancer predict prognosis and immunotherapy outcomes. J Immunother Cancer. 2021 Nov;9(11):e003214. doi: 10.1136/jitc-2021-003214. PMID 34795005
- [Derived] Chen X, Wu X, Wu H, Gu Y, Shao Y, Shao Q, Zhu F, Li X, Qian X, Hu J, Zhao F, Mao W, Sun J, Wang J, Han G, Li C, Xia Y, Seesaha PK, Zhu D, Li H, Zhang J, Wang G, Wang X, Li X, Shu Y. Camrelizumab plus gemcitabine and oxaliplatin (GEMOX) in patients with advanced biliary tract cancer: a single-arm, open-label, phase II trial. J Immunother Cancer. 2020 Nov;8(2):e001240. doi: 10.1136/jitc-2020-001240. PMID 33172881